CLINICAL TRIAL: NCT05370976
Title: Efficacy and Safety of Cytotect®CP, Hyperimmune Anti-CMV IVIg as CMV Prophylaxis in Patients Developing Acute Grade II-IV GVHD After Allogeneic Hematopoietic Cell Transplantation: A Prospective, Open-label, Phase II Study
Brief Title: Efficacy and Safety of Cytotect®CP, Hyperimmune Anti-CMV IVIg as CMV Prophylaxis in Patients Developing Acute Grade II-IV GVHD After Allogeneic Hematopoietic Cell Transplantation.
Acronym: CMV-GVHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inclusion difficulties
Sponsor: University Hospital, Lille (Other)
Collaborators: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020_42; 2020-004698-30 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-05-19; First posted 2022-05-12 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Drug: Cytotect®CP

INTERVENTIONS:
Drug: Cytotect®CP — Cytotect®CP in two phases:
  Induction phase: 1 ml/kg/week for 4 weeks Maintenance phase: 1 ml/kg/2 weeks for 12 weeks or corticosteroid dose < 0.5 mg/kg, according to which condition occurs first.
  Patients developing CMV infection under Cytotect®CP must be given standard anti-CMV treatment (Gancyclovir or Foscarnet) according to their center procedure. Cytotect®CP will be maintained

SUMMARY:
Many risk factors are known to be associated with high risk of developing CMV infection in positive CMV-serostatus patients: negative CMV-serostatus donor, unrelated or mismatched donor, use of antithymocyte globulin (ATG), and development of GVHD. Acute GVHD occurs during the first hundred days after transplantation. In spite of systematic GVHD prophylactic using immunosuppressive agents, approximately 50% of transplantation recipients develop GVHD. The first-line treatment of acute GVHD is methylprednisolone 2 mg/kg/day. Probably because of the use corticosteroids but also due to the GVHD itself, approximately 46% of CMV seropositive patients develop CMV infection (report from the national database of the SFGM-TC, data unpublished yet).

CMV infection leads to longer duration of hospitalization and increases the risk of mortality, particularly in cases of CMV disease. Available antiviral agents used to prevent CMV infections are generally reputed to cause significant side effects. These agents can prevent full immunological post-transplant reconstitution and cause profound cytopenia. Some agents may be responsible for renal impairment, which prevents continuation of immunosuppressive treatment; this is especially the case with calcineurin inhibitors in allo-HCT patients. Indeed, compared to placebo, intravenous ganciclovir has been shown to reduce the risk of CMV infection and disease, although it did not appear to improve overall survival. However, it was responsible for 30% of cases of severe neutropenia in allo-HCT patients, increasing the risk of bacterial and fungal coinfections. CMV infection treatment is commonly based on ganciclovir and foscavir and, to a lesser extent, on other drugs, including cidofovir. However, these drugs cause high levels of toxicity, resulting in myelotoxicity in the case of ganciclovir, or, in the case of foscavir and cidofovir, potential renal failure, incurring treatment discontinuation.

CMV prophylaxis using drugs with fewer side-effects is necessary in patients at high risk of CMV infection.

With its safety profile, Cytotect®CP offers an alternative option for CMV prophylaxis with avoidance of renal and bone marrow impairment.

Considering the high risk of developing CMV infection, we decided to investigate the efficacy and safety of Cytotect®CP in patients requiring systematic corticosteroids (≥ 1 mg/kg/day) for an initial episode of grade II-IV acute GVHD following a first allo-HCT.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Patients before day from 29 days to 150 days of first allo-HCT
* Any indication, any stem cell source, any conditioning, any donor type or HLA-matching
* Patients with positive CMV-serostatus before transplant
* Patients with first episode of grade II-IV acute GVHD requiring systemic corticosteroids ≥1 mg/kg/day
* Absence of CMV infection at the time of inclusion
* Absence of other viral infections (EBV, adenovirus, BK virus) at the time of inclusion
* Absence of dialysis
* Absence of thrombotic microangiopathy
* Absence of macrophage activation syndrome

Exclusion Criteria:

* - Patients receiving corticosteroids > 0.5 mg/kg/day for more than 5 days before inclusion
* Uncontrolled CMV infection within 02 weeks before inclusion
* Inability to understand the investigational nature of the study or to give informed consent
* ECOG Performance Status ≥ 3
* Evidence of relapse of underlying disease
* Patients receiving or having received anti-CMV treatment within 30 days before inclusion (acyclovir and valacyclovir are not considered as CMV prophylaxis)
* Hypersensitivity to Cytotect®CP or to any of the excipients
* Hypersensitivity to human immunoglobulins, especially in patients with antibodies against IgA
* Patients with any contra-indication to Cytotect®CP
* Females either pregnant/breast-feeding or planning to become pregnant
* Patients developing post-DLI grade II-IV acute GVHD
* Freedom privacy
* Absence of medical insurance cover

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Rate of CMV infection within 16 weeks of Cytotect®CP therapy. | within 16 weeks

SECONDARY OUTCOMES:
Time from inclusion to death from any cause or death without relapse of the underlying disease within 6 months | from inclusion to 16 weeks
Time from inclusion to EBV, adenovirus or BK virus co-infection ≤ 16 weeks. | within the 16 weeks from inclusion
Time from inclusion to CMV infection ≤ 16 weeks. | within the 16 weeks from inclusion
Time from inclusion to CMV disease ≤ 16 weeks | within the 16 weeks from inclusion
Frequency of adverse events (grades 3 and 4) | from 1st administration of Cytotect®CP throughout the 4 weeks after the last administration of Cytotect®CP, an average 20 weeks
Analysis of immune reconstitution under Cytotect®CP. | Througth study completion, an average 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Yakoub-Agha, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France